CLINICAL TRIAL: NCT04227288
Title: An Investigator Initiated Study Evaluating the Efficacy and Tolerability of Enstilar Foam (Calcipotriene and Betamethasone Dipropionate) in Patients With Nail Psoriasis
Brief Title: A Study Evaluating the Efficacy and Tolerability of Enstilar Foam in Patients With Nail Psoriasis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: LEO Pharma (Industry)
Responsible Party: Principal Investigator, Boni Elewski, Primary Investigator, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300003797
Record Dates: First submitted 2019-11-26; First posted 2020-01-13 (Actual); Results first posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Nail Psoriasis
Keywords: Enstilar Foam
MeSH Terms: interventions — betamethasone dipropionate, calcipotriol drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Enstilar Foam (Experimental): Eligible subjects will be provided once daily Enstilar Foam (calcipotriene and betamethasone dipropionate).
  Interventions: Drug: Enstilar Foam

INTERVENTIONS:
Drug: Enstilar Foam — Subjects will be instructed to apply a thin layer on the nail plate, around the nail plate and under the nail plate. The patient will be instructed to apply one application at night immediately before bed and not wash their hands before morning. All subjects who completed the 6-month treatment will be followed for 1 month after discontinuation.
  Other Names: calcipotriene and betamethasone dipropionate

SUMMARY:
The aim of the study is to evaluate the efficacy and safety of Enstilar Foam (calcipotriene and betamethasone dipropionate) for the treatment of nail psoriasis.

DETAILED DESCRIPTION:
Eligible subjects will be provided once daily Enstilar Foam (calcipotriene and betamethasone dipropionate). Subjects will be instructed to apply a thin layer on the nail plate, around the nail plate and under the nail plate. The subject will be instructed to apply one application at night immediately before bed and not wash their hands before morning. All subjects who completed the 6-month treatment will be followed for 1 month after discontinuation.

ELIGIBILITY:
Inclusion Criteria:

* Must have a diagnosis of nail psoriasis in fingernail or toenails
* History of plaque psoriasis or psoriatic arthritis
* Target nail will be KOH negative for dermatophyte fungus
* Must give written informed consent prior to study procedures being conducted, also give consent to the release and use of protected health information (PHI)
* Between the ages of 18 and 85 years old
* Candidate for topical therapy in the opinion of the investigator

Exclusion Criteria:

* Males and Females unable to practice effective contraception throughout the study
* Unable to comply with the protocol
* Nursing mothers, pregnant women, and women planning to become pregnant while in this study
* Patients with erythrodermic or pustular psoriasis
* Sustained treatment to target fingernail within 6 months prior to screening
* History of trauma or surgery to target fingernail
* History of disease known to affect nails such as lichen planus, onychomycosis
* History of systemic psoriasis therapy for less than 6 months

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boni E Elewski, Dr, Principal Investigator — University of Alabama at Birmingham/Dermatology
Locations (1):
- The University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Enstilar Foam: Open-label drug administration group. No comparator.
  Enstilar foam
Period: Overall Study
Arm/Group | Enstilar Foam
Started | 6
Completed | 3
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Enstilar Foam
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 2
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Clinical Improvement in Nail Thickness of Target Nail at Week 24 Compared to Baseline.
Description: The target nail will be defined as the nail that has the highest nail thickness score at baseline. This nail will remain the target nail for the remainder of the study. Number of participants achieving clinical improvement as measure by the nail thickness (hyperkeratosis) measurement at week 24 compared to baseline.
Time Frame: 24 Weeks
Measure: Number; unit: Participants who experienced improvement
Units Other Than Participants: Fingernail
Arm/Group | Enstilar Foam
Number analyzed (Participants) | 3
Number analyzed (Fingernail) | 3
Participants who experienced improvement | 2

2. Secondary Outcome: Modified mNAPSI (Modified Nail Area Psoriasis Severity Index) Score of Fingernails at Week 24 Compared to Baseline
Description: All fingernails will be analyzed for the outcome measure. mNAPSI is an objective scoring system administered by trained healthcare providers. The range of possible scores is 0 to 130, with a score of 0 indicating absence of nail disease and a score of 130 indicating the most severe nail disease. A decrease in mNAPSI score indicates improvement. The mNAPSI 75 response is defined as at least 75% reduction from baseline in mNAPSI
Time Frame: 24 weeks
Population: All fingernails for each participant were analyzed at week 24 only.
Measure: Number; unit: Fingernails
Units Other Than Participants: Fingernails
Arm/Group | Enstilar Foam
Number analyzed (Participants) | 3
Number analyzed (Fingernails) | 30
Fingernails | 18

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over the entirety of the study, 28 weeks for each participant.
Arm/Group | Enstilar Foam
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 2/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enstilar Foam (N=6)
Torn Bicep (Musculoskeletal and connective tissue disorders) | 1 (1)
Torn Rotator Cuff (Musculoskeletal and connective tissue disorders) | 1 (1)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2017-08-22): https://cdn.clinicaltrials.gov/large-docs/88/NCT04227288/Prot_001.pdf